CLINICAL TRIAL: NCT00122473
Title: Open-label Trial of Glivec® (Imatinib Mesylate) in Patients With Primary or Recurrent Dermatofibrosarcoma Protuberans
Brief Title: Imatinib in Dermatofibrosarcoma Protuberans (DFSP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dermatologic Cooperative Oncology Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADO/VOD DFSP 001; CSTI571BDE25
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Dermatofibrosarcoma
Keywords: Dermatofibrosarcoma; Imatinib; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Dermatofibrosarcoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib (Glivec)

SUMMARY:
The purpose of this study is to determine whether imatinib is effective in the treatment of primary and recurrent dermatofibrosarcoma protuberans (DFSP).

DETAILED DESCRIPTION:
This study is aimed to investigate the efficacy of imatinib (Glivec) in the treatment of primary and locally relapsed dermatofibrosarcoma protuberans (DFSP). DFSP is a cutaneous neoplasm well known for its overexpression of the platelet-derived growth factor (PDGF). Herein, imatinib provides a systemic treatment option that offers the possibility of a reduction of the wide surgical margins used today in surgery of primary DFSP, or even of a complete avoidance of surgical treatment in this disease. Since imatinib exerts its function via interference with protein tyrosine kinase activities, it inhibits the platelet-derived growth factor receptor (PDGF-R) signaling cascade that plays a crucial role in the pathogenesis and tumor growth of DFSP. Since imatinib has been shown to shrink metastatic lesions of DFSP, there is a strong rationale to expect that it also decreases cell proliferation and tumor growth in primary DFSP.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary or recurrent dermatofibrosarcoma protuberans
* Measurable tumor parameters (by magnetic resonance imaging [MRI])
* Patient >/= 18 years of age
* ECOG performance status < 3
* Adequate organ function
* Patients must be able to swallow capsules
* Female patients of childbearing potential must have negative pregnancy test
* Written, voluntary, informed consent; must include investigational use of tumor tissue biopsies.

Exclusion Criteria:

* Any evidence of distant metastases
* Patient has received any other investigational agents within 28 days of first day of study drug dosing
* Patient is < 5 years free of another primary malignancy except basal cell skin cancer or cervical carcinoma in situ
* Grade III/IV cardiac problems as defined by the New York Heart Association
* Severe and/or uncontrolled medical disease
* Known diagnosis of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2007-01

PRIMARY OUTCOMES:
Tumor response at 6 and 12 weeks

SECONDARY OUTCOMES:
Rate of relapse within the first 2 years
Association of tumor response with cytogenetic and receptor expression status

CONTACTS AND LOCATIONS:
Overall Officials: Selma Ugurel, MD, Principal Investigator — Skin Cancer Unit, German Cancer Research Center Heidelberg and Department of Dermatology, University Hospital of Mannheim, Mannheim, Germany; Dirk Schadendorf, MD, Principal Investigator — Skin Cancer Unit, German Cancer Research Center Heidelberg and Department of Dermatology, University Hospital of Mannheim, Mannheim, Germany
Locations (4):
- Germany (4):
  - Skin Cancer Unit, German Cancer Research Center and Department of Dermatology, University Hospital of Mannheim, Mannheim, Baden-Wurttemberg
  - Department of Dermatology, ElbeKliniken - Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Department of Dermatology, The Saarland University Hospital, Homburg/Saar, Saarland
  - Department of Dermatology, Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt

REFERENCES:
- [Background] McArthur GA, Demetri GD, van Oosterom A, Heinrich MC, Debiec-Rychter M, Corless CL, Nikolova Z, Dimitrijevic S, Fletcher JA. Molecular and clinical analysis of locally advanced dermatofibrosarcoma protuberans treated with imatinib: Imatinib Target Exploration Consortium Study B2225. J Clin Oncol. 2005 Feb 1;23(4):866-73. doi: 10.1200/JCO.2005.07.088. PMID 15681532
- [Background] Labropoulos SV, Fletcher JA, Oliveira AM, Papadopoulos S, Razis ED. Sustained complete remission of metastatic dermatofibrosarcoma protuberans with imatinib mesylate. Anticancer Drugs. 2005 Apr;16(4):461-6. doi: 10.1097/00001813-200504000-00014. PMID 15746584
- [Background] Price VE, Fletcher JA, Zielenska M, Cole W, Viero S, Manson DE, Stuart M, Pappo AS. Imatinib mesylate: an attractive alternative in young children with large, surgically challenging dermatofibrosarcoma protuberans. Pediatr Blood Cancer. 2005 May;44(5):511-5. doi: 10.1002/pbc.20249. PMID 15503291
- [Background] Mizutani K, Tamada Y, Hara K, Tsuzuki T, Saeki H, Tamaki K, Matsumoto Y. Imatinib mesylate inhibits the growth of metastatic lung lesions in a patient with dermatofibrosarcoma protuberans. Br J Dermatol. 2004 Jul;151(1):235-7. doi: 10.1111/j.1365-2133.2004.06024.x. No abstract available. PMID 15270901
- [Background] McArthur G. Molecularly targeted treatment for dermatofibrosarcoma protuberans. Semin Oncol. 2004 Apr;31(2 Suppl 6):30-6. doi: 10.1053/j.seminoncol.2004.03.038. PMID 15176002
- [Background] Sirvent N, Maire G, Pedeutour F. Genetics of dermatofibrosarcoma protuberans family of tumors: from ring chromosomes to tyrosine kinase inhibitor treatment. Genes Chromosomes Cancer. 2003 May;37(1):1-19. doi: 10.1002/gcc.10202. PMID 12661001
- [Background] Maki RG, Awan RA, Dixon RH, Jhanwar S, Antonescu CR. Differential sensitivity to imatinib of 2 patients with metastatic sarcoma arising from dermatofibrosarcoma protuberans. Int J Cancer. 2002 Aug 20;100(6):623-6. doi: 10.1002/ijc.10535. PMID 12209598
- [Background] Rubin BP, Schuetze SM, Eary JF, Norwood TH, Mirza S, Conrad EU, Bruckner JD. Molecular targeting of platelet-derived growth factor B by imatinib mesylate in a patient with metastatic dermatofibrosarcoma protuberans. J Clin Oncol. 2002 Sep 1;20(17):3586-91. doi: 10.1200/JCO.2002.01.027. PMID 12202658
- [Background] Sjoblom T, Shimizu A, O'Brien KP, Pietras K, Dal Cin P, Buchdunger E, Dumanski JP, Ostman A, Heldin CH. Growth inhibition of dermatofibrosarcoma protuberans tumors by the platelet-derived growth factor receptor antagonist STI571 through induction of apoptosis. Cancer Res. 2001 Aug 1;61(15):5778-83. PMID 11479215
- [Background] Greco A, Roccato E, Miranda C, Cleris L, Formelli F, Pierotti MA. Growth-inhibitory effect of STI571 on cells transformed by the COL1A1/PDGFB rearrangement. Int J Cancer. 2001 May 1;92(3):354-60. doi: 10.1002/ijc.1190. PMID 11291071
- [Background] Shimizu A, O'Brien KP, Sjoblom T, Pietras K, Buchdunger E, Collins VP, Heldin CH, Dumanski JP, Ostman A. The dermatofibrosarcoma protuberans-associated collagen type Ialpha1/platelet-derived growth factor (PDGF) B-chain fusion gene generates a transforming protein that is processed to functional PDGF-BB. Cancer Res. 1999 Aug 1;59(15):3719-23. PMID 10446987